CLINICAL TRIAL: NCT00251940
Title: A 24-Week Randomised, Double-Blind, Parallel-Group, Multi-Centre, Placebo-Controlled Study to Evaluate the Efficacy, Safety and Tolerability of Tesaglitazar Therapy When Added to the Therapy of Patients With Type 2 Diabetes Poorly Controlled on Sulphonylurea Alone
Brief Title: GALLANT 7 Tesaglitazar Add-on to Sulphonylurea
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The development program has been terminated
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D6160C00032; EudraCT No 2004-001144-71
Record Dates: First submitted 2005-11-09; First posted 2005-11-11 (Estimated); Last update posted 2008-03-17 (Estimated); Status verified 2008-03

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

INTERVENTIONS:
Drug: Tesaglitazar 0.5 or 1 mg
Drug: Glibenclamide 2.5, 5, 10 or 15 mg

SUMMARY:
This is a 24-week randomized double-blind, parallel-group, multi-center, placebo-controlled study of tesaglitazar (0.5 mg and 1 mg) given as add-on therapy to sulphonylurea in patients with type 2 diabetes, not adequately controlled on optimized sulphonylurea treatment and on diet/lifestyle advice during the titration and run-in period. The study comprises a 2-week enrollment period, 6 week placebo metformin titration period, 2-week single-blind run-in period, followed by a 24-week double blind treatment period and a 3-week follow-up period

ELIGIBILITY:
Inclusion Criteria:

* Provision of a written informed consent
* Female patients: postmenopausal, hysterectomized, or if of childbearing potential, using a reliable method of birth control
* Diagnosed with type 2 diabetes
* Treated with diet alone or treatment with a single oral antidiabetic agent or low doses of two oral antidiabetic agents

Exclusion Criteria:

* Type 1 diabetes
* New York Heart Association heart failure Class III or IV
* Treatment with chronic insulin
* History of hypersensitivity or intolerance to any peroxisome proliferator-activated receptor agonist (like Actos or Avandia), fenofibrate, metformin or 3-hydroxy-3-methylglutaryl coenzyme A reductase inhibitor (statin)
* History of drug-induced myopathy or drug-induced creatine kinase elevation, liver enzyme elevations, neutropenia (low white blood cells)
* Creatinine levels above twice the normal range
* Creatine kinase above 3 times the upper limit of normal
* Received any investigational product in other clinical studies within 12 weeks
* Any clinically significant abnormality identified on physical examination, laboratory tests or electrocardiogram, which in the judgment of the investigator would compromise the patient's safety or successful participation in the clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 555
Dates: Start 2004-07; Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Absolute change from baseline to end of randomized treatment period in glycosylated hemoglobin A1c (HbA1c)

SECONDARY OUTCOMES:
Changes in the following variables from baseline to the end of the randomized treatment period:
• The change in fasting plasma glucose (FPG), insulin, proinsulin and C-peptide
• Insulin sensitivity by assessment of change in the calculated variable homeostasis assessment model
• Lipid parameters (triglyceride [TG], total cholesterol, high-density lipoprotein cholesterol [HDL C], non-HDL C, low-density lipoprotein cholesterol [LDL C], apolipoproteins [Apo] A-I, Apo B, Apo CIII, free fatty acids, lipoprotein particle size and c
• C-reactive protein, LDL C/HDL C ratio and Apo B/Apo A-I ratio
• FPG, homeostasis assessment model, insulin, proinsulin, C-peptide
• Tumor necrosis factor-alpha, intracellular adhesion molecule-1
• Fibrinogen
• Urinary albumin excretion
• Waist/hip ratio
• Responder analyses for HbA1c, FPG, TG, HDL C, total cholesterol, non HDL C and LDL C according to pre-specified values
• Proportion of patients reaching pre-specified target levels for HbA1c, FPG, TG, HDL C, non-HDL C and LDL C
• Pharmacokinetics of tesaglitazar
• Safety and tolerability of tesaglitazar by assessment of adverse events, laboratory values, electrocardiogram, pulse, blood pressure, hypoglycemic events, body weight, cardiac evaluation, and physical examination

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Galida Medical Science Director, MD, Study Director — AstraZeneca
Locations (84):
- Australia (8):
  - Research Site, Adelaide
  - Research Site, Brisbane
  - Research Site, Cairns
  - Research Site, Geelong
  - Research Site, Melbourne
  - Research Site, Perth
  - Research Site, Sydney
  - Research Site, Tasmania
- France (13):
  - Research Site, Angers
  - Research Site, Hyères
  - Research Site, La Garde
  - Research Site, La Seyne-sur-Mer
  - Research Site, Laval
  - Research Site, Le Brusc
  - Research Site, Le Lavandou
  - Research Site, Montrevault
  - Research Site, Paris
  - Research Site, Saint-Cyr
  - Research Site, Six-Fours-les-Plages
  - Research Site, Tiercé
  - Research Site, Toulon
- Israel (8):
  - Research Site, Ashkelon
  - Research Site, Haifa
  - Research Site, Holon
  - Research Site, Jerusalem
  - Research Site, Rishon LeZiyyon
  - Research Site, Safed
  - Research Site, Tel Aviv
  - Research Site, Tel Litwinsky
- Norway (16):
  - Research Site, Bergen
  - Research Site, Elverum
  - Research Site, Enebakk
  - Research Site, Fredrikstad
  - Research Site, Gamle Fredrikstad
  - Research Site, Hamar
  - Research Site, Haugesund
  - Research Site, Hurdal
  - Research Site, Inderøy
  - Research Site, Lena
  - Research Site, Levanger
  - Research Site, Oslo
  - Research Site, Rud
  - Research Site, Sedsmokorset
  - Research Site, Soerumsand
  - Research Site, Stavanger
- Philippines (3):
  - Research Site, Manila
  - Research Site, Marikina City
  - Research Site, Pasig
- South Africa (4):
  - Research Site, Cape Town
  - Research Site, Chatsworth
  - Research Site, Gauteng
  - Research Site, Pretoria
- South Korea (2):
  - Research Site, Seoul
  - Research Site, Suwon
- Spain (7):
  - Research Site, Alzira (Valencia)
  - Research Site, Barcelona
  - Research Site, Guissona (Lleida)
  - Research Site, Madrid
  - Research Site, San Sebastian de Los Reyes ( Madrid)
  - Research Site, San Vicente de Raspeig (Alicante)
  - Research Site, Valencia
- United Kingdom (21):
  - Research Site, Dublin, Ireland
  - Research Site, Aberdeen
  - Research Site, Barnsley
  - Research Site, Bath
  - Research Site, Belfast
  - Research Site, Birmingham
  - Research Site, Cardiff
  - Research Site, Coventry
  - Research Site, Dundee
  - Research Site, East Sussex
  - Research Site, Edinburgh
  - Research Site, Glasgow
  - Research Site, Leeds
  - Research Site, Liverpool
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Shrewsbury
  - Research Site, Surrey
  - Research Site, West Midlands
  - Research Site, Wiltshire
  - Research Site, Wrexham
- Vietnam (2):
  - Research Site, Hanoi
  - Research Site, Ho Chi Minh City